CLINICAL TRIAL: NCT02288572
Title: Mechanisms of Action of Probiotic and Protective Bacteria PCS 20, PCS 26, and LGG in Prevention of the Metabolic Syndrome
Brief Title: Probiotic Bacteria in Prevention of the Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Maribor (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Mario Gorenjak, Biomedical field scientist, University Maribor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MGPS001
Record Dates: First submitted 2014-11-02; First posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Metabolic Syndrome X
Keywords: metabolic syndrome X; obesity; insulin resistance; dyslipidemia; probiotic bacteria
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Insulin Resistance; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactobacillus plantarum PCS 26 (Active Comparator): Dosage: 1.000.000.000 Colony Forming Units (CFU) per day in powdery form for 3 months Vehicle: 70 % glucose, 15 % powder milk, 15 % whey
  Interventions: Dietary Supplement: Lactobacillus plantarum PCS 26
- Placebo (Placebo Comparator): Only vehicle components in powdery form for 3 months Vehicle: 70 % glucose, 15 % powder milk, 15 % whey
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum PCS 26 — Taking dietary supplement on a daily basis which corresponds to 1.000.000.000 CFU of Lactobacillus plantarum PCS 26 per day for 3 months.
  Arms: Lactobacillus plantarum PCS 26
Dietary Supplement: Placebo — Taking dietary supplement on a daily basis for 3 months.
  Arms: Placebo

SUMMARY:
The metabolic syndrome is increasing worldwide, including developing countries. The metabolic syndrome is composed of clinical expressed symptoms as central obesity, high blood pressure, raised fasting plasma glucose or diagnosed diabetes, low HDL, and raised serum triglycerides. All those components together or independently contribute to the development of cardiovascular diseases, which are the leading cause of death in the modern world. The results from previous studies have shown that probiotic bacteria have an influence on health improvement, and can exert positive effects on diseases as diabetes, high blood pressure, dyslipidemia and low-grade inflammation, which are all components of the metabolic syndrome. The objectives of this study were to investigate which of probiotic strains Lactobacillus plantarum PCS 20, Lactobacillus plantarum PCS 26 in Lactobacillus rhamnosus GG exert positive effects in the cascade of molecular reactions at the level of small intestines, at remodeling of monocytes/macrophages and adipocytes in human cell model of non-cancerous origin, and to provide scientific explanation of mechanisms of possible multi-leveled activity of selected probiotic strains in patients with metabolic syndrome. For this purpose, the investigators divided this research into two parts. The first part consisted of pre-clinical in-vitro laboratory study. It examined the mechanisms of actions of probiotic cultures with the use of functional cell models of non-cancerous origin, more specifically, with the use of cell lines of human intestinal epithelium, human monocytes/macrophages and human visceral preadipocytes. In in-vitro laboratory study, the investigators demonstrated that probiotic strain Lactobacillus plantarum PCS 26 exerts positive effects, which could help to relieve the particular components of the syndrome in the host with metabolic syndrome. The second part of the research consisted of prospective, double-blind and placebo-controlled in-vivo pilot clinical study, which included 16 volunteers with the metabolic syndrome. Results have shown that probiotic strain Lactobacillus plantarum PCS 26 exerts positive effects on reduction of waist circumference, on lowering of serum cholesterol concentration, and on maintenance of serum adiponectin levels. Those effects together can contribute to the alleviation of the metabolic syndrome, especially in terms of clinical manifestation and risks in relation to cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* visceral obesity and at least two of other components: raised fasting serum glucose or known diabetes type 2; raised fasting serum triglycerides; raised fasting serum cholesterol; raised fasting serum LDL and low fasting serum HDL; high blood pressure, more than 130/85 mmHg.

Exclusion Criteria:

* planned invasive procedure or surgery (whole body);
* planned surgery in mouth cavity;
* weakened immune system or taking immunosuppressives;
* diagnosed inflammatory bowel disease;
* known or diagnosed lactose intolerance.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Serum lipids concentrations after daily consumption of dietary supplement in patients with the metabolic syndrome | 3 months
  Serum total cholesterol, triglycerides, LDL and HDL concentrations

SECONDARY OUTCOMES:
Measures of body composition after daily consumption of dietary supplement in patients with the metabolic syndrome | 3 months
  Body weight, body mass without body fat, total body fat, body volume, muscle mass, body mass index, visceral fat, subcutaneous fat, blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Skok, DSc, MD, Study Chair — University Medical Centre Maribor; Mario Gorenjak, DSc, MBioinf, BHSc, Principal Investigator — Faculty of Medicine, University of Maribor